CLINICAL TRIAL: NCT06890390
Title: TSPO PET in the Evaluation of Neuroinflammation in Patients with Multiple System Atrophy
Status: Recruiting | Type: Observational
Sponsor: Min Zhao,MD (Other)
Responsible Party: Sponsor-Investigator, Min Zhao,MD, Doctor, Central South University
Organization: Central South University (Other)
Other Study IDs: Rapid24280
Record Dates: First submitted 2025-03-20; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-04

CONDITIONS: Multiple System Atrophy - Cerebellar Subtype (MSA-C); Multiple System Atrophy - Parkinsonian Subtype (MSA-P)
Keywords: Multiple System Atrophy; PETCT; TSPO
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MSA-C group: Clinically confirmed MSA and clinically probable MSA according to the 2022 MDS MSA diagnostic criteria，and have symptoms of MSA-C type (with cerebellar ataxia as the main manifestation) mainly include progressive cerebellar ataxia and autonomic dysfunction.
- MSA-P group: Clinically confirmed MSA and clinically probable MSA according to the 2022 MDS MSA diagnostic criteria，and have symptoms of MSA-P (multiple system atrophy-P type) mainly include autonomic dysfunction, Parkinson's syndrome and cerebellar ataxia.
- healthy control group: The healthy person who age, gender and other basic conditions matched with the MSA cohort population，and voluntarily participate in this study and sign the informed consent.

SUMMARY:
The aim of this study was to apply PET/MR techniques targeting TSPO to explore the temporal and spatial alterations characterizing neuroinflammation in MSA patients, and to assess its value as a biomarker for diagnostic typing, disease severity, and prognosis of MSA disease.

ELIGIBILITY:
Inclusion Criteria:

* Age> 35 years old, gender is not limited;
* Clinically confirmed MSA and clinically probable MSA according to the 2022 MDS MSA diagnostic criteria;
* all patients had been ruled out of polyQ disease by genetic testing;
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* pregnancy or breastfeeding;
* contraindications to MRI examination or inability to cooperate in completing neuroimaging examination;
* previous history of other neurological disorders or presence of other organic intracranial lesions on neuroimaging that cannot be interpreted by MSA, such as epilepsy, trauma, tumors, or high-grade cerebral white matter degeneration (Fazekas grade 2 and above);
* History of alcohol or drug abuse

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who came to Third Xiangya Hospital of Central South University for consultation or online questionnaire recruitment
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value ratio(SUVR) | From enrollment to the end of treatment at 4 weeks

SECONDARY OUTCOMES:
UMSARS | From enrollment to the end of treatment at 4 weeks
  Unified Multiple System Atrophy Rating Scale
H-Y stage | From enrollment to the end of treatment at 4 weeks
SCOPA-AUT | From enrollment to the end of treatment at 4 weeks
  Parkinson's Disease Autonomic Symptoms Scale
Wexner score | From enrollment to the end of treatment at 4 weeks
  Wexner Continence Grading Scale
Frontal Assessment Battery | From enrollment to the end of treatment at 4 weeks
MoCA score | From enrollment to the end of treatment at 4 weeks
  Montreal Cognitive Assessment
TSPO Single nucleotide polymorphism genotyping | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Third Xiangya Hospital of Central South University, Hunan, Changsha, China

IPD SHARING:
Plan to Share IPD: Yes